CLINICAL TRIAL: NCT03040492
Title: Vitamin D Receptor Polymorphisms and Non-Melanoma Skin Cancer Risks in Alabama Population
Brief Title: Vitamin D Receptor Polymorphisms and Non-Melanoma Skin Cancer Risk
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Nabiha Yusuf, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: X120713008
Record Dates: First submitted 2017-01-27; First posted 2017-02-02 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Skin Cancer, Non-Melanoma
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — Biospecimens retained for further analysis of polymorphisms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to discover whether certain Vitamin D Receptor (VDR) gene polymorphisms are associated with an increased risk of cutaneous basal cell carcinoma (BCC) and/or cutaneous squamous cell carcinoma (SCC) in an Alabama population. Participant demographic information such as physical characteristics (e.g., ethnicity), family history, and cancer diagnosis will be collected in order to determine if there are relationships between the gene polymorphisms, cancer diagnosis, and these characteristics.

DETAILED DESCRIPTION:
The purpose of this study is to discover whether certain Vitamin D Receptor (VDR) gene polymorphisms are associated with an increased risk of cutaneous basal cell carcinoma (BCC) and/or cutaneous squamous cell carcinoma (SCC) in an Alabama population. Participant demographic information such as physical characteristics (e.g., ethnicity), family history, and cancer diagnosis will be collected in order to determine if there are relationships between the gene polymorphisms, cancer diagnosis, and these characteristics. By identifying the VDR polymorphisms for the Apa1, Taq1, Bsm1, and Fok1 genes within the participant population and comparing the genotypes to controls, the investigators hope to demonstrate which gene polymorphisms indicate an increased risk for SCC or BCC.

Inclusion- patients with a non-melanoma skin cancer. Participants must be 50 years old or older. Controls- patients without non-melanoma skin cancer and who have no family history of skin cancer. They must also be 50 years old or older; Inclusion for both groups- English speakers and patients at the Kirklin Clinic during the months of our data collection. Exclusion criteria will be patients younger than 50 years old or who have a diagnosis of melanoma or other type of cancer, or who are non-English speakers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-melanoma skin cancer (cases)
* Patients without non-melanoma skin cancer or history of non-melanoma skin cancer (controls)
* Age 50 and older
* Native English speakers
* Patients at Kirklin Clinic

Exclusion Criteria:

* Age less than 50
* Diagnosis of melanoma or other type of cancer
* Non-English speakers

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patient group consisted of 100 subjects with a BCC or SCC diagnosis, visiting the Dermatology Clinics at The Kirklin Clinic at the University of Alabama at Birmingham between 2012 and 2014
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-10-31 (Actual); Primary Completion 2013-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
SIngle nucleotide polymorphisms (SNP) | 2 years
  Number of patients with the presence or absence of VDR SNP in their DNA isolated from their blood samples. PCR will be performed on the DNA samples for using specific primers for SNP, and the PCR products will be sequenced for detection of SNP.

CONTACTS AND LOCATIONS:
Locations (1):
- The Kirklin Clinic, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No